CLINICAL TRIAL: NCT00411515
Title: A Prospective Randomized Trial on Mycophenolate Mofetil in Risk Penetrating Keratoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FR-2000-05-2006-06
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Corneal Transplantation

INTERVENTIONS:
Drug: Mycophenolate Mofetil 2x 1g

SUMMARY:
The purpose of this prospectively randomized multicentre study was to prove the efficacy and safety of mycophenolate mofetil (MMF) to preventing graft rejection and improvement of clear graft survival following high-risk keratoplasty.

The patients of the MMF group receive MMF orally 2x1 g daily for 6 months. Endpoints were immune reaction free and clear graft survival and the occurence of side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Keratoplasty with increased risk for immunologic graft rejection in the abscence of other risk factors for graft failure. (repeat keratoplasty, steroid-response, limbo-keratoplasty, oversized graft.

Exclusion Criteria:

* Normal risk cases. Herpes-Keratitis. Glaucoma. Limbus stem cell deficiency.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reinhard, Prof. MD, Study Chair — University Eye Hospital, Freiburg
Locations (1):
- University Eye hospital, Freiburg im Breisgau, Germany

REFERENCES:
- [Result] Reinhard T, Mayweg S, Sokolovska Y, Seitz B, Mittelviefhaus H, Engelmann K, Voiculescu A, Godehardt E, Sundmacher R. Systemic mycophenolate mofetil avoids immune reactions in penetrating high-risk keratoplasty: preliminary results of an ongoing prospectively randomized multicentre study. Transpl Int. 2005 Jun;18(6):703-8. doi: 10.1111/j.1432-2277.2005.00126.x. PMID 15910297
- [Derived] Birnbaum F, Mayweg S, Reis A, Bohringer D, Seitz B, Engelmann K, Messmer EM, Reinhard T. Mycophenolate mofetil (MMF) following penetrating high-risk keratoplasty: long-term results of a prospective, randomised, multicentre study. Eye (Lond). 2009 Nov;23(11):2063-70. doi: 10.1038/eye.2008.402. Epub 2009 Jan 16. PMID 19151659